CLINICAL TRIAL: NCT05281471
Title: A Randomized Phase 3 Study Assessing the Efficacy and Safety of Olvi-Vec Followed by Platinum-doublet Chemotherapy and Bevacizumab Compared With Physician's Choice of Chemotherapy and Bevacizumab in Women With Platinum-Resistant/Refractory Ovarian Cancer (PRROC) (OnPrime, GOG-3076)
Brief Title: Efficacy & Safety of Olvi-Vec and Platinum-doublet + Bevacizumab Compared to Physician's Choice of Chemotherapy and Bevacizumab in Platinum-Resistant/Refractory Ovarian Cancer (PRROC) (OnPrime, GOG-3076)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genelux Corporation (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Olvi-Vec-022; GOG-3076 (Other: GOG Foundation)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Platinum-resistant Ovarian Cancer; Platinum-refractory Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; High-grade Serous Ovarian Cancer; Endometrioid Ovarian Cancer; Ovarian Clear Cell Carcinoma
Keywords: olvimulogene nanivacirepvec; GL-ONC1; GLV-1h68; oncolytic virus; virotherapy; viral therapy; immunotherapy; immunochemotherapy; combination therapy; vaccinia virus; ovarian cancer; fallopian tube cancer; primary peritoneal cancer; platinum resistant; platinum refractory; recurrent ovarian cancer; platinum resensitization; chemoresistance; heavily pre-treated; immune activation; reversal of platinum resistance or refractoriness; resensitize
MeSH Terms: conditions — Fallopian Tube Neoplasms; Vaccinia; Ovarian Neoplasms | interventions — Cisplatin; taxane; Paclitaxel; Docetaxel; 130-nm albumin-bound paclitaxel; liposomal doxorubicin; Bevacizumab; Biosimilar Pharmaceuticals

STUDY DESIGN:
Intervention Model Description: Randomization (2:1) is either into the Experimental Arm which is Olvi-Vec followed by platinum-doublet chemotherapy and bevacizumab or into the Active Comparator Arm which is Physician's Choice of chemotherapy and bevacizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olvi-Vec + Platinum-doublet & bevacizumab (Experimental): Olvi-Vec: A total of 2 consecutive days of intraperitoneal catheter infusions in Week 0
  Platinum-doublet & bevacizumab (or biosimilar) administered beginning in Week 4 (preferred), but no later than Week 5
  Interventions: Biological: olvimulogene nanivacirepvec; Drug: Platinum chemotherapy: carboplatin (preferred) or cisplatin; Drug: Non-platinum chemotherapy: Physician's Choice of gemcitabine, taxane (paclitaxel, docetaxel or nab-paclitaxel) or pegylated liposomal doxorubicin; Drug: Bevacizumab (or biosimilar)
- Physician's Choice of Chemotherapy & bevacizumab (Active Comparator): Physician's Choice of chemotherapy & bevacizumab (or biosimilar) administered beginning in Week 0. Physician's Choice of chemotherapy includes either a single agent non-platinum chemotherapy, or as platinum chemotherapy is allowed as an option, a platinum-doublet (i.e., platinum agent combined with a non-platinum agent).
  Interventions: Drug: Platinum chemotherapy: carboplatin (preferred) or cisplatin; Drug: Non-platinum chemotherapy: Physician's Choice of gemcitabine, taxane (paclitaxel, docetaxel or nab-paclitaxel) or pegylated liposomal doxorubicin; Drug: Bevacizumab (or biosimilar)

INTERVENTIONS:
Biological: olvimulogene nanivacirepvec — Olvi-Vec is an engineered oncolytic vaccinia virus
  Other Names: GL-ONC1 and GLV-1h68
  Arms: Olvi-Vec + Platinum-doublet & bevacizumab
Drug: Platinum chemotherapy: carboplatin (preferred) or cisplatin — Administered according to local practice
Drug: Non-platinum chemotherapy: Physician's Choice of gemcitabine, taxane (paclitaxel, docetaxel or nab-paclitaxel) or pegylated liposomal doxorubicin — Administered according to local practice
Drug: Bevacizumab (or biosimilar) — Administered according to local practice

SUMMARY:
The OnPrime study is a multi-center, randomized open-label phase 3 study evaluating the safety and efficacy of Olvi-Vec followed by platinum-doublet chemotherapy and bevacizumab compared to the Active Comparator Arm with Physician's Choice of chemotherapy and bevacizumab in women diagnosed with platinum-resistant/refractory ovarian cancer (includes fallopian tube cancer and primary peritoneal cancer). This Phase III trial builds on the efficacy and safety data reported in the previous Phase II VIRO-15 trial with promising objective response rate and progression-free survival observed in heavily pre-treated patients with platinum-resistant/refractory ovarian cancer. The phase II results also showed that the intra-peritoneal route of delivery was efficient in generating tumor cell killing and immune activation, and led to clinical reversal of platinum-resistance or refractoriness in this difficult-to-treat patient population.

DETAILED DESCRIPTION:
Olvi-Vec (olvimulogene nanivacirepvec, aka GL-ONC1, laboratory name: GLV-1h68) is an oncolytic vaccinia virus-based immunotherapy. This study is to test the hypothesis that the combination of Olvi-Vec followed by further chemotherapy is particularly effective against established tumors by virus-mediated immune activation and re-sensitization of tumor cells to chemotherapy. Participant population includes histologically confirmed non-resectable platinum-resistant/refractory ovarian cancer (PRROC). Determination of progression-free survival, safety and overall survival are key objectives. Participants randomized into the Experimental Arm will receive a single-cycle (2 infusions on two consecutive days) of Olvi-Vec through an intraperitoneal catheter. The catheter is then removed, and patients receive systemically administered platinum-doublet chemotherapy and bevacizumab. The control arm receives the Physician's Choice of chemotherapy and bevacizumab at the same dose and schedule. Biological samples will be obtained from some Experimental Arm participants for virus-shedding testing. Assessment of response to treatment in both arms will be by RECIST 1.1 and iRECIST as assessed by Blinded Independent Central Review. Maintenance/continued treatment with non-platinum chemotherapy and bevacizumab is dependent on a participant being clinically stable until confirmed progressive disease by iRECIST or can no longer tolerate therapy.

Dr. Robert W. Holloway (AdventHealth Cancer Institute, Orlando, FL) will serve as the National Principal Investigator for this Phase 3 study in PRROC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed (from prior treatment) non-resectable ovarian, fallopian tube or primary peritoneal cancer.
* High-grade serous [including malignant mixed Mullerian tumor (MMMT) with metastasis that contains high-grade epithelial carcinoma, FIGO grades 2 & 3 allowed], endometrioid, or clear-cell ovarian cancer.
* Performance status ECOG of 0 or 1.
* Life expectancy of at least 6 months.
* Received a minimum of 3 prior lines (including the 1st line) of systemic therapy with no maximal limit.
* Platinum-resistant or -refractory disease based on platinum-free interval (PFI) from the last dose of the most recent. platinum-based line of therapy (must have received a minimum of 2 doses of platinum in that line) to subsequent disease progression based on radiological assessment. Platinum-refractory: PFI of < 1 month (including disease progression while on platinum-based therapy). Platinum-resistant: PFI of 1-6 months.
* Received prior bevacizumab (or biosimilar) treatment.
* No contraindication to receive carboplatin, cisplatin or bevacizumab (or biosimilar).
* Have disease progression after last prior line of therapy based on radiological assessment prior to randomization.
* At least 1 measurable target lesion per RECIST 1.1 based on abdominal/pelvis imaging scan at screening.
* Evidence by CT and/or PET scans or physical exam of abdominal/pelvis region likely having disease in the peritoneal cavity (i.e., peritoneal carcinomatosis).
* Adequate renal, hepatic, bone marrow function, adequate coagulation tests, adequate immune function by lymphocyte count.

Exclusion Criteria:

* Tumors of mucinous, low-grade serous, squamous cell, small cell neuroendocrine subtypes, MMMT tumors absent an epithelial component on recent biopsy, or non-epithelial ovarian cancers (e.g., germ cell tumors, Sex-cord tumors).
* Bowel obstruction within last 3 months prior to screening.
* Active urinary tract infection, pneumonia, other systemic infections.
* Active gastrointestinal bleeding.
* Known current central nervous system (CNS) metastasis.
* Inflammatory diseases of the bowel.
* History of HIV infection.
* Active hepatitis B virus or hepatitis C virus within 4 weeks prior to study.
* History of thromboembolic event within the prior 3 months.
* Contraindications for intraperitoneal (IP) catheter placement: Bowel obstruction with distended abdomen, rigid abdomen with bulky anterior wall carcinomatosis, abdominal wall hernia mesh that precludes laparoscopic entry to abdomen.
* Clinically significant cardiac disease at screening (New York Heart Association Class III/IV).
* Acute cerebrovascular event(s) such as cerebrovascular accident (CVA) or transient ischemic attack (TIA) in previous 6 months.
* Oxygen saturation <90%.
* Received prior virus-based gene therapy or therapy with cytolytic virus of any type.
* Receiving concurrent antiviral agent.
* Prior malignancy of other histology active within previous 3 years except for locally curable cancers apparently cured such as basal/squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of cervix or breast, any other stage I/II local malignancies.
* Received chemotherapy, radiotherapy, other anti-cancer biologic therapies within 4 weeks prior to planned treatment.
* Underwent surgery within 4 weeks, or have insufficient recovery from surgical-related trauma or wound healing, prior to first study treatment in either Arm.
* Receiving immunosuppressive therapy or steroids (except acute concurrent corticosteroid of no more than 20 mg per day for medical management with prednisolone equivalent.
* Symptomatic malignant ascites or pleural effusions defined as rapidly progressive ascites with abdominal distension and gastrointestinal dysfunction, pleural effusions with respiratory difficulties requiring frequent paracentesis > once every 14 days.
* Known hypersensitivity to gentamicin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by RECIST 1.1 in the Intention-to-Treat (ITT) population (all randomized participants regardless of whether they received any dose of treatment) | From date of randomization up to 12 months
  To assess progression-free survival from time of randomization until first documented disease progression based on radiological assessment or death from any cause.

SECONDARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events in the ITT population | From date of first study treatment until death or study completion; assessed up to 36 months
  Determine safety and tolerability of administering multiple doses of Olvi-Vec via intraperitoneal catheter in combination with platinum-doublet and bevacizumab (or biosimilar) as assessed by CTCAE v. 5.0 following initiation of study treatment until end of study participation.
Duration of Response (DOR) by RECIST 1.1 in the ITT population | From date of randomization up to 12 months
  Time from date of first response until the first date of progressive disease based on radiological assessment.
PFS by RECIST 1.1 in the modified ITT (mITT) population (participants who received at least 1 dose of treatment in either Arm) | From date of randomization up to 12 months
  Time from randomization to first documented disease progression based on radiological assessment or death from any cause.
PFS by iRECIST in the ITT population | From date of randomization up to 12 months
  Time from randomization to first documented disease progression with confirmatory imaging scan performed 4-8 weeks after unconfirmed disease progression or death from any cause.
Overall Response Rate (ORR) by RECIST 1.1 in the ITT population | From date of randomization up to 12 months
  Ratio of the sum of CR & PR divided by the number of ITT participants from start of treatment to confirmation of response.
Overall Survival in the ITT population | From date of randomization until death or study completion; assessed up to 36 months
  Time from randomization until date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Holloway, MD, Principal Investigator — AdventHealth Cancer Institute
Locations (31):
- United States (31):
  - The University of South Alabama, Mitchell Cancer Institute, Mobile, Alabama
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - UC San Diego Health - Moores Cancer Center, La Jolla, California
  - Hoag Gynecologic Oncology, Newport Beach, California
  - UCI Health Chao Family Comprehensive Cancer Center, Orange, California
  - AdventHealth Cancer Institute, Orlando, Florida
  - Sarasota Memorial Research Institute, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Holy Cross Hospital, Silver Spring, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope, Reno, Nevada
  - Stony Brook Cancer Center, Stony Brook, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Kettering Health, Kettering, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Oklahoma University Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - AHN West Penn Hospital, Pittsburgh, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Erlanger Health, Inc., Chattanooga, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Science Center at Houston, McGovern Medical School, Houston, Texas
  - Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mori KM, Giuliano PD, Lopez KL, King MM, Bohart R, Goldstein BH. Pronounced clinical response following the oncolytic vaccinia virus GL-ONC1 and chemotherapy in a heavily pretreated ovarian cancer patient. Anticancer Drugs. 2019 Nov;30(10):1064-1066. doi: 10.1097/CAD.0000000000000836. PMID 31567308
- [Result] Manyam M, Stephens AJ, Kennard JA, LeBlanc J, Ahmad S, Kendrick JE, Holloway RW. A phase 1b study of intraperitoneal oncolytic viral immunotherapy in platinum-resistant or refractory ovarian cancer. Gynecol Oncol. 2021 Dec;163(3):481-489. doi: 10.1016/j.ygyno.2021.10.069. Epub 2021 Oct 20. PMID 34686353
- [Result] Holloway RW, Mendivil AA, Kendrick JE, Abaid LN, Brown JV, Fitzsimmons CK, Kennard JA, King M, LeBlanc J, Lopez K, Manyam M, McKenzie ND, Mori KM, Stephens AJ, Sarfraz A. 2020 International Gynecologic Cancer Society, Oral Plenary Session presentation of VIRO-15 Phase 2 Trial Data, Robert Holloway, AdventHealth Cancer Institute, Orlando, FL. International Journal of Gynecologic Cancer 2020;30:A9-A10
- [Result] Holloway RW, Mendivil AA, Kendrick JE, Abaid LN, Brown JV, LeBlanc J, McKenzie ND, Mori KM, Ahmad S. Clinical Activity of Olvimulogene Nanivacirepvec-Primed Immunochemotherapy in Heavily Pretreated Patients With Platinum-Resistant or Platinum-Refractory Ovarian Cancer: The Nonrandomized Phase 2 VIRO-15 Clinical Trial. JAMA Oncol. 2023 Jul 1;9(7):903-908. doi: 10.1001/jamaoncol.2023.1007. PMID 37227734
- [Derived] Holloway RW, Thaker P, Mendivil AA, Ahmad S, Al-Niaimi AN, Barter J, Beck T, Chambers SK, Coleman RL, Crafton SM, Crane E, Ramez E, Ghamande S, Graybill W, Herzog T, Indermaur MD, John VS, Landrum L, Lim PC, Lucci JA, McHale M, Monk BJ, Moore KN, Morris R, O'Malley DM, Reid TJ, Richardson D, Rose PG, Scalici JM, Silasi DA, Tewari K, Wang EW. A phase III, multicenter, randomized study of olvimulogene nanivacirepvec followed by platinum-doublet chemotherapy and bevacizumab compared with platinum-doublet chemotherapy and bevacizumab in women with platinum-resistant/refractory ovarian cancer. Int J Gynecol Cancer. 2023 Sep 4;33(9):1458-1463. doi: 10.1136/ijgc-2023-004812. PMID 37666539
- See also: Genelux Corporation's Sponsor website — http://www.genelux.com/
- See also: Genelux Corporation's preclinical publications — https://www.genelux.com/pre-clinical-publications/
- See also: Genelux Corporation's clinical publications — http://www.genelux.com/clinical-publications/
- See also: The GOG Foundation's Partner website — http://www.gog.org